CLINICAL TRIAL: NCT00059904
Title: An Open-Labeled, Phase II Study of Rituximab in Combination With Recombinant IL-2 for Relapsed or Refractory Non-Hodgkin's Lymphoma of Intermediate- or High-Grade Histology
Brief Title: Rituximab and Interleukin-2 in Treating Patients With Relapsed or Refractory Intermediate- or High-Grade Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CHIR-IL2005-A01; MSKCC-03004; CDR0000298986 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-05-06; First posted 2003-05-07 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2004-07

CONDITIONS: Lymphoma
Keywords: recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult immunoblastic large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic | interventions — aldesleukin; Rituximab

INTERVENTIONS:
Biological: aldesleukin
Biological: rituximab

SUMMARY:
RATIONALE: Monoclonal antibodies such as rituximab can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Interleukin-2 may stimulate a person's white blood cells to kill cancer cells. Combining rituximab with interleukin-2 may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combining rituximab with interleukin-2 in treating patients who have relapsed or refractory intermediate- or high-grade non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the clinical efficacy of rituximab and interleukin-2 in patients with relapsed or refractory intermediate- or high-grade non-Hodgkin's lymphoma.
* Determine the 2-year progression-free survival of patients treated with this regimen.
* Determine the safety of this regimen in these patients.
* Correlate response with natural killer cell numbers and rituximab, interleukin-2 (IL-2), and soluble IL-2 receptor levels in patients treated with this regimen.

OUTLINE: This is an open-label, multicenter study.

Patients receive rituximab IV once weekly on weeks 1-4 and interleukin-2 subcutaneously 3 times weekly on weeks 2-9. Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed every 12 weeks for 2 years.

PROJECTED ACCRUAL: A total of 50-100 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of intermediate- or high-grade non-Hodgkin's lymphoma according to the Working Formulation, including the following subtypes:

  * Diffuse large cell lymphoma
  * Diffuse mixed cell lymphoma
  * Immunoblastic large cell lymphoma
* CD20+ disease
* Measurable progressive or refractory disease
* No primary CNS lymphoma or lymphomatous meningitis NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Lymphocyte count less than 20,000/mm^3
* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 75,000/mm^3
* Hemoglobin at least 9.5 g/dL

Hepatic

* SGOT and SGPT no greater than 1.5 times upper limit of normal
* Bilirubin normal
* No liver disease
* Hepatitis C-seropositive patients are allowed provided they have no active disease, as demonstrated by any of the following:

  * Undetectable hepatitis C viral loads
  * Biopsy showing no active disease
  * Normal transaminases on at least 3 different occasions within the past year

Renal

* Creatinine normal

Cardiovascular

* No clinically significant cardiac dysfunction
* No myocardial infarction within the past 6 months
* No heart failure within the past 6 months

Pulmonary

* No clinically significant pulmonary dysfunction
* Patients with prior radiotherapy to the lung or autologous transplantation must have FEV greater than 50% and DLCO greater than 50% within 8 weeks before study treatment

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No significant infections within the past 2 weeks (including pneumonia or bronchitis)
* No history of autoimmune disease
* No prior or concurrent malignancy except inactive nonmelanoma skin cancer, carcinoma in situ of the cervix, or other solid tumor curatively treated with no evidence of recurrence within the past 2 years
* No symptomatic thyroid disease requiring medical intervention other than replacement treatment for hypothyroidism
* No prior type 1 hypersensitivity or anaphylactic reactions to murine products, rituximab, or radioimmunoconjugated anti-CD20 antibody infusion

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 3 months since prior autologous bone marrow transplantation
* No prior allogeneic bone marrow transplantation
* No prior interleukin-2
* No prior interferon (alfa, beta, or gamma)
* No concurrent basiliximab, daclizumab, or monoclonal antibody OKT3

Chemotherapy

* More than 30 days since prior chemotherapy
* No concurrent anticancer chemotherapy

Endocrine therapy

* More than 2 weeks since prior systemic steroids
* No concurrent systemic corticosteroids

Radiotherapy

* More than 30 days since prior radiotherapy
* No concurrent radiotherapy

Surgery

* More than 30 days since prior major surgery

Other

* More than 30 days since other prior investigational drugs
* More than 30 days since prior immunosuppressive medications
* No concurrent immunosuppressive medications including the following:

  * Cyclosporine
  * Mycophenolate mofetil
  * Tacrolimus
  * Sirolimus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-01; Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tarun Kewalramani, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States